CLINICAL TRIAL: NCT04321161
Title: Analysis of T Cell Metabolism and Immune Phenotype in Relapsed Acute Myeloid Leukemia Patients Receiving Donor Lymphocyte Infusions and Bicanorm (Sodium Bicarbonate)
Brief Title: Analysis of T Cell Metabolism in Relapsed AML Patients With DLIs and Bicanorm Treatment
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Freiburg (Other)
Responsible Party: Principal Investigator, Robert Zeiser, Director of the Division of Tumor Immunology, University of Freiburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BICARB_AMLrelapse
Record Dates: First submitted 2020-03-20; First posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Acute Myeloid Leukemia, in Relapse
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AML relapse under DLI and Bicanorm treatment (Experimental): Analysis of T cell metabolism, immune phenotype and serum pH before and after Bicanorm (Sodium bicarbonate) treatment.
  Interventions: Drug: Bicanorm

INTERVENTIONS:
Drug: Bicanorm — Treatment of patients with relapsed AML after allo-HCT receiving DLIs with Bicanorm (1-1-1) for 7 days.
  sodium hydrogen carbonate (1 g per 1 tablet) = sodium ion (11,9 mmol per 1 tablet) = sodium ion (273 mg per 1 tablet) = hydrogen carbonate ion (11,9 mmol per 1 tablet)
  Other Names: Sodium bicarbonate

SUMMARY:
In this study, the outcomes of relapsed AML patients receiving DLIs and Bicanorm (Sodium bicarbonate) were analyzed including T cell metabolism and immune phenotype.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) patients suffering from relapse after allogeneic hematopoietic cell transplantation (allo-HCT) have a poor survival outcome. Donor lymphocyte infusions (DLIs) to induce graft-versus-leukemia (GvL) effects have a limited survival benefit.

Extensive preclinical studies have shown a beneficial effect of sodium bicarbonate on metabolic fitness of leukemia-reactive T cells in GvL AML models. Therefore, the investigators aimed to investigate a potential benefit of Bicanorm (Sodium bicarbonate) treatment accompanying DLIs in relapsed AML patients. The investigators determined the metabolic and immune phenotype of T cells isolated from patients receiving DLIs before and after Bicanorm (Sodium bicarbonate) treatment.

ELIGIBILITY:
Inclusion Criteria:

* confirmed AML relapse after allo-HCT
* patients receiving DLIs
* age ≥ 18 years
* written informed consent
* ability to understand the nature of the study and the study related procedures and to comply with them

Exclusion Criteria:

* age < 18 years
* lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
T cell glycolytic activity | 2 months
  Extracellular acidification rate (ECAR) determined by live-cell metabolic assay using the Seahorse Analyzer
T cell respiratory activity | 2 months
  Oxygen consumption rate (OCR) determined by live-cell metabolic assay using the Seahorse Analyzer
T cell phenotype | 2 months
  T cell cytokine and effector molecule production determined by flow cytometric analysis

SECONDARY OUTCOMES:
Serum pH | 2 months
  Measurement of serum pH

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zeiser, Prof. Dr., Principal Investigator — Medical Center University of Freiburg
Locations (1):
- Medical Center University of Freiburg, Freiburg im Breisgau, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang CH, Qiu J, O'Sullivan D, Buck MD, Noguchi T, Curtis JD, Chen Q, Gindin M, Gubin MM, van der Windt GJ, Tonc E, Schreiber RD, Pearce EJ, Pearce EL. Metabolic Competition in the Tumor Microenvironment Is a Driver of Cancer Progression. Cell. 2015 Sep 10;162(6):1229-41. doi: 10.1016/j.cell.2015.08.016. Epub 2015 Aug 27. PMID 26321679
- [Background] Pilon-Thomas S, Kodumudi KN, El-Kenawi AE, Russell S, Weber AM, Luddy K, Damaghi M, Wojtkowiak JW, Mule JJ, Ibrahim-Hashim A, Gillies RJ. Neutralization of Tumor Acidity Improves Antitumor Responses to Immunotherapy. Cancer Res. 2016 Mar 15;76(6):1381-90. doi: 10.1158/0008-5472.CAN-15-1743. Epub 2015 Dec 30. PMID 26719539
- [Background] Schmid C, Labopin M, Nagler A, Bornhauser M, Finke J, Fassas A, Volin L, Gurman G, Maertens J, Bordigoni P, Holler E, Ehninger G, Polge E, Gorin NC, Kolb HJ, Rocha V; EBMT Acute Leukemia Working Party. Donor lymphocyte infusion in the treatment of first hematological relapse after allogeneic stem-cell transplantation in adults with acute myeloid leukemia: a retrospective risk factors analysis and comparison with other strategies by the EBMT Acute Leukemia Working Party. J Clin Oncol. 2007 Nov 1;25(31):4938-45. doi: 10.1200/JCO.2007.11.6053. Epub 2007 Oct 1. PMID 17909197